CLINICAL TRIAL: NCT05438966
Title: Body Composition and Dietary Intake Status of Adult Slovenes After the Covid-19 Epidemic
Brief Title: Nutritional Status of Adult Slovenes After the Covid-19 Epidemic
Acronym: SloFitCovid
Status: Completed | Type: Observational
Sponsor: Barbara Jakše s.p. (Other)
Responsible Party: Principal Investigator, Boštjan Jakše, Boštjan Jakše, Principal Investigator, Barbara Jakše s.p.
Other Study IDs: KR6
Record Dates: First submitted 2022-06-28; First posted 2022-06-30 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Body Weight; Nutrition, Healthy; COVID-19 Pandemic
MeSH Terms: conditions — Body Weight; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
There is objective need to examine nutritional status (i.e., body mass index (BMI), body composition and dietary intake) of healthy adult Slovenes after SARS-CoV-2 (Covid-19) epidemic period.

In the Slovenian (pair of European Union) adult population (with only 2 million inhabitants), we do not yet have representative data on the body composition of adult Slovenes published in the scientific literature.

In the study after the Covid-19 pandemic period (4th wave) the investigators will use medically approved body analyzer (Tanita 780 S MA, Tokyo, Japan) and standardized food frequency questionnaire (FFQ). In addition, the investigators will measured body height of the participants with a portable altimeter (ADE MZ10042, Germany).

The research will include randomly recruited adults (participants) who will attend various free or/and paid publicly available seminars, congresses and fairs in Slovenia, directly unrelated topics to physical activity or healthy eating (i.e., healthy and active lifestyle) thus obtaining a more realistic current population status.

DETAILED DESCRIPTION:
In the study investigators will randomly but voluntarily enroll 700-1000 healthy adult participants within inclusion/exclusion criteria that are willing to participate in the study. Investigators anticipate that for this number of adults (aged 18-80 years) will require approx. 5000 invited candidates (10-15 events), of both sexes.

The methods to be used are body composition monitor and FFQ. In addition to the assessment of BMI and body composition status, we will compare the proportion of obese subjects according to BMI and body fat percentage threshold criteria (by World Health Organization). For the dietary intake analysis the investigators will use the national a dietary software program, OPEN Platform for Clinical Nutrition, which is a web-based application developed by the Jožef Stefan Institute in Slovenia.

The power of the sample was calculated on the basis of published body composition data on the adult population of the scientific monographs of the Slovenian National Institute of Public Health and data on the BMI of the scientific research on the dietary intake status of adults (SI.Menu).

The participants included in the study will signed consent form for inclusion in the study and will not be remunerated financially for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* No BMI restriction
* Randomly invited

Exclusion Criteria:

* Without currently competitive or top level athletes
* Without pregnant or lactating women and physically handicapped individuals
* Without active common chronic diseases (i.e., cancer, CVD, autoimmune diseases ect.)
* Without individuals with a pacemaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult Slovenes
Sampling Method: Probability Sample
Enrollment: 833 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Body weight status | June-September 2022
  Body weight measured with medically approved body composition monitor
Height status | June-September 2022
  Height status measured with medically approved weighing scale with height rod
Body mass index (BMI) status | June-September 2022
  Measured body weight and body height will be combined to report BMI in kg/m2
Body fat percentege status | June-September 2022
  Body fat percentage measured with medically approved body composition monitor
Muscle mass percantage status | June-September 2022
  Muscle mass percantage measured with medically approved body composition monitor

SECONDARY OUTCOMES:
Dietary intake status | June-September 2022
  Dietary intake measured by standardized food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Boštjan Jakše, PhD, Principal Investigator — Independent Researcher; Stanislav Pinter, PhD, Study Chair — University of Ljubljana
Locations (1):
- Faculty of sport, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pravst I, Lavrisa Z, Hribar M, Hristov H, Kvarantan N, Seljak BK, Gregoric M, Blaznik U, Gregoric N, Zaletel K, Oblak A, Osredkar J, Zmitek K, Kusar A. Dietary Intake of Folate and Assessment of the Folate Deficiency Prevalence in Slovenia Using Serum Biomarkers. Nutrients. 2021 Oct 28;13(11):3860. doi: 10.3390/nu13113860. PMID 34836112
- [Background] Clarys P, Deliens T, Huybrechts I, Deriemaeker P, Vanaelst B, De Keyzer W, Hebbelinck M, Mullie P. Comparison of nutritional quality of the vegan, vegetarian, semi-vegetarian, pesco-vegetarian and omnivorous diet. Nutrients. 2014 Mar 24;6(3):1318-32. doi: 10.3390/nu6031318. PMID 24667136
- [Background] De Keyzer W, Dekkers A, Van Vlaslaer V, Ottevaere C, Van Oyen H, De Henauw S, Huybrechts I. Relative validity of a short qualitative food frequency questionnaire for use in food consumption surveys. Eur J Public Health. 2013 Oct;23(5):737-42. doi: 10.1093/eurpub/cks096. Epub 2012 Jul 26. PMID 22843611
- [Background] Korosec M, Golob T, Bertoncelj J, Stibilj V, Seljak BK. The Slovenian food composition database. Food Chem. 2013 Oct 1;140(3):495-9. doi: 10.1016/j.foodchem.2013.01.005. Epub 2013 Jan 17. PMID 23601397
- [Background] Verney J, Schwartz C, Amiche S, Pereira B, Thivel D. Comparisons of a Multi-Frequency Bioelectrical Impedance Analysis to the Dual-Energy X-Ray Absorptiometry Scan in Healthy Young Adults Depending on their Physical Activity Level. J Hum Kinet. 2015 Oct 14;47:73-80. doi: 10.1515/hukin-2015-0063. eCollection 2015 Sep 29. PMID 26557191